CLINICAL TRIAL: NCT02891083
Title: Multi-center Prospective Randomized Controlled Clinical Trial of Postoperative Adjuvant Chemotherapy, Adjuvant Radiotherapy, or Surgery Alone for High-risk Histological Node Negative Patients With Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Adjuvant Therapies or Surgery Alone for High Risk pN0 Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Sun Yat-sen University (Other); Sichuan Cancer Hospital and Research Institute (Other); Hunan Cancer Hospital (Other); Fujian Cancer Hospital (Other Government); Fudan University (Other); Qingdao University (Other); Fujian Medical University (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Wentao Fang, Chief Director,Clinical Center of Esophageal Diseases,Shanghai Jiao tong University, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016shchest
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Esophageal Neoplasms
Keywords: adjuvant chemotherapy; adjuvant radiotherapy; lymph node metastasis; surgery; squamous cell carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Lymphatic Metastasis; Carcinoma, Squamous Cell | interventions — Chemotherapy, Adjuvant; Paclitaxel; Cisplatin; TP protocol; Radiotherapy, Adjuvant; Cobalt-60; Control Groups; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adjuvant chemotherapy group (Experimental): Surgery followed by adjuvant chemotherapy,with Paclitaxel and Cisplatin.
  Interventions: Drug: Adjuvant chemotherapy (Paclitaxel and Cisplatin)
- Adjuvant radiotherapy group (Experimental): Surgery followed by 50Gy adjuvant radiotherapy
  Interventions: Radiation: Adjuvant radiotherapy
- Control group (Other): Surgery alone
  Interventions: Other: Control group (Surgery alone)

INTERVENTIONS:
Drug: Adjuvant chemotherapy (Paclitaxel and Cisplatin) — Adjuvant chemotherapy group: three cycles: (Paclitaxel: 175mg/m2 ivgtt, 3h, d1 4week × 3 and cisplatin: 75mg/m2 ivgtt, d1 4 week × 3)
  Other Names: Paclitaxel and Cisplatin
  Arms: Adjuvant chemotherapy group
Radiation: Adjuvant radiotherapy — Target: the upper mediastinum and bilateral supraclavicular region (Upper bound: thyrocricoid, lower bound: carina of 3cm)
  Dose: 50Gy
  Technology: strong tone
  Segmentation: conventional segmentation 2Gy/d
  Other Names: cobalt-60
  Arms: Adjuvant radiotherapy group
Other: Control group (Surgery alone)
  Other Names: Surgery alone
  Arms: Control group

SUMMARY:
Histological Node Negative thoracic esophageal squamous cell carcinoma（pN0 ESCC） after radical resection still carries the risk of recurrence after complete surgical resection, especially in some high-risk patients. There are still lack of knowledge on postoperative treatment indication and methods for pN0 ESCC.Our previous study has shown that risk of recurrence is associated with the location and cell differentiation of primary tumor, as well as the presence of lymphovascular invasion. This project is designed to study the efficacy of adjuvant therapies for at patients with pN0 ESCC and above mentioned risk factors of recurrence after radical surgery. We aim to compare the differences among adjuvant chemotherapy, adjuvant radiotherapy, and surgery alone for pN0 ESCC by prospective randomized controlled trial. There has been no similar studies in esophageal cancer previously reported with similar design. The results of this study is expected to have a high clinical relevance.

DETAILED DESCRIPTION:
The study is designed to be a prospective randomized controlled trial, aiming to compare the impact of adjuvant chemotherapy with Paclitaxel and Cisplatin, adjuvant radiotherapy with IMRT of 50Gy, and surgery alone on the disease free survival (DFS) of patients with high-risk pN0 thoracic esophageal squamous cell carcinoma. Pathological staging is to be based on the 7th UICC edition, after radical resection and systemic lymph node dissection,for accurate staging.Patients with pT1b-T4a disease, proved to be pN0 upon pathological examination, meet at least one of the risk factors in the inclusion criteria, and without any exclusion criteria are to be randomized into one of the three study arms.Definition of high-risk factors for recurrence include: (1)Tumor location: in the middle or upper third thoracic esophagus; (2) Presence of LVI or submucosal metastasis; (3) Cell differentiation: poorly differentiated or undifferentiated.

Primary endpoint:

To observe and compare Disease-Free Survivals (DFS) among the three study arms.

Secondary endpoint:

To observe and compare Overall Survivals (OS) among the three study arms, and to compare adverse events between adjuvant chemotherapy and adjuvant radiation groups.

Additional instructions:

No.

ELIGIBILITY:
Inclusion Criteria:

1. Patient: No pretreatment before surgery.Informed consent signed after screening;
2. Surgery: Complete (R0) resection of tumor, with thoraco- abdominal two-field or cervico-thoraco-abdominal three-field lymph node dissection through transthoracic esophagectomy. At least 12 stations and 12 lymph nodes should be harvested, including bilateral recurrent laryngeal nerve nodes. Both open thoracotomy and minimally invasive thoracoscopic/laparoscopic approaches are allowed and histopathological examination confirmed the diagnosis of the patients with at least cleaning more or equal to 12 stations and 12 lymph nodes;
3. Histology: Thoracic esophageal squamous cell carcinoma, with no nodal involvement (pN0) after pathological examination;
4. Staging: Tumor T stage T1b-T4a according to the 7th UICC esophageal cancer staging system;
5. Definition of high risk for recurrence: meet at least one of the three below.

   A: Primary tumor located in middle or upper third of thoracic esophagus

   B: Presence of lymphovascular invasion (LVI) or submucosal metastasis

   C: Cell differentiation:Low grade or undifferentiated
6. Performance status: ECOG score 0-2;
7. Cardiac function:NYHA classification 1-2. Normal electrocardiogram;
8. Renal function: Normal serum creatinine level (SCr = 120mol/L) and creatinine clearance rate (CCr = 60 ml/min);
9. Hepatic function: Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) level less than or equal to 2.0 times the upper limit of normal (ULN). Serum alkaline phosphatase (ALP) level less than or equal to four times the upper limit of normal value. Serum total bilirubin level less than or equal to 1.5 times the upper limit of the normal value;
10. Hematopoietic function: White blood cell count (WBC) equal to or more than 4000 / μL,neutrophils (ANC) absolute count is more than or equal to 1500 / μ L, platelet count more than or equal to 100000/ μ L, hemoglobin equal to or more than 10.0 g / dl.

Exclusion Criteria:

1. Surgery through Left thoracic or transhiatal approach, whereby complete lymphadenectomy is not achieved;
2. Patients experienced severe postoperative complication and thus, are unable to tolerate any adjuvant therapy;
3. Patients who have concommitant other malignant tumor;
4. Patients with abnormal coagulation function, with bleeding tendencies (such as active peptic ulcer) or are currently receiving thrombolysis or anticoagulation therapies;
5. Severe cardiac comorbidities, including congestive heart failure,uncontrolled cardiac arrhythmia, unstable angina pectoris, myocardial infarction within six months,severe heart valve disease, or intractable hypertension;
6. Severe hepatic or renal insufficiency;
7. Poor mental status or mental disorders, poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years
side effect of adjuvant therapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wentao Fang, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guo XF, Mao T, Gu ZT, Ji CY, Fang WT, Chen WH. Clinical study on postoperative recurrence in patients with pN0 esophageal squamous cell carcinoma. J Cardiothorac Surg. 2014 Aug 28;9:150. doi: 10.1186/s13019-014-0150-4. PMID 25164541
- [Result] Shim YM, Kim HK, Kim K. Comparison of survival and recurrence pattern between two-field and three-field lymph node dissections for upper thoracic esophageal squamous cell carcinoma. J Thorac Oncol. 2010 May;5(5):707-12. doi: 10.1097/JTO.0b013e3181d3ccb2. PMID 20421764
- [Result] Ando N, Iizuka T, Ide H, Ishida K, Shinoda M, Nishimaki T, Takiyama W, Watanabe H, Isono K, Aoyama N, Makuuchi H, Tanaka O, Yamana H, Ikeuchi S, Kabuto T, Nagai K, Shimada Y, Kinjo Y, Fukuda H; Japan Clinical Oncology Group. Surgery plus chemotherapy compared with surgery alone for localized squamous cell carcinoma of the thoracic esophagus: a Japan Clinical Oncology Group Study--JCOG9204. J Clin Oncol. 2003 Dec 15;21(24):4592-6. doi: 10.1200/JCO.2003.12.095. PMID 14673047
- [Result] Tachimori Y, Nagai Y, Kanamori N, Hokamura N, Igaki H. Pattern of lymph node metastases of esophageal squamous cell carcinoma based on the anatomical lymphatic drainage system. Dis Esophagus. 2011 Jan;24(1):33-8. doi: 10.1111/j.1442-2050.2010.01086.x. PMID 20626450
- [Result] Wu SG, Dai MM, He ZY, Sun JY, Lin HX, Lin H, Li Q. Patterns of Regional Lymph Node Recurrence After Radical Surgery for Thoracic Esophageal Squamous Cell Carcinoma. Ann Thorac Surg. 2016 Feb;101(2):551-7. doi: 10.1016/j.athoracsur.2015.08.057. Epub 2015 Oct 31. PMID 26530541